CLINICAL TRIAL: NCT01027663
Title: Impact of Host Iron Status and Iron Supplement Use on Growth and Viability of the Erythrocytic Stage of Plasmodium Falciparum
Brief Title: Impact of Host Iron Status and Iron Supplement Use on Erythrocytic Stage of Plasmodium Falciparum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Raj Kasthuri, MD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-0559
Record Dates: First submitted 2009-12-04; First posted 2009-12-09 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Iron Deficiency Anemia; Malaria
Keywords: anemia; malaria
MeSH Terms: conditions — Anemia, Iron-Deficiency; Malaria; Anemia | interventions — Iron-Dextran Complex; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Iron Deficiency Anemia (No Intervention)
- Hereditary Hemochromatosis (No Intervention)
- Iron Supplements (Active Comparator)
  Interventions: Dietary Supplement: Iron Supplement

INTERVENTIONS:
Dietary Supplement: Iron Supplement — Iron supplementation (325 mg of ferrous sulfate) once daily for the 2 month duration of the study.
  Other Names: Ferrous sulfate
  Arms: Iron Supplements

SUMMARY:
The purpose of this study is to perform laboratory based studies to determine if the growth and development of the malaria parasite is effected by iron status of its host (the person infected with the malaria parasite). Iron deficiency affects over 500 million people including many pregnant women and children from areas of the world that are plagued by malaria. Some population based studies have suggested that iron deficiency protects people from getting malaria and this has raised questions about the wisdom of public health policies that provide universal iron supplementation in countries where malaria is common. We will use red blood cells and sera from patients with iron deficiency anemia, hereditary hemochromatosis and normal individuals who are taking iron supplements to look at this question in a very systematic way. This study should provide information for or against a possible mechanism by which iron deficiency may affect the malaria parasite. The results will contribute to efforts to develop evidence-based public health policies on iron supplementation policies in malaria-endemic areas.

There are three different types of individuals involved in this study (1) people with iron deficiency anemia who will be taking iron supplementation (2) people without iron deficiency anemia who will be taking iron supplementation and (3) people with a condition called hereditary hemochromatosis who have an excess of iron in their bodies.

DETAILED DESCRIPTION:
Purpose: This proposal is aimed at studying the effect of an individual's iron status and iron supplementation on the growth and viability of the malarial parasite Plasmodium falciparum. The overall goal is to provide evidence to support the development of evidence-based programs to improve global health policy on iron supplementation in areas of the world with high malaria transmission. Current WHO recommendations include routine supplementation of women and children. Recently however, the wisdom of this policy when applied to areas afflicted with high rates of malaria has come under scrutiny. This proposal will study the effects of red blood cells (RBCs) and sera from iron overloaded patients (with hereditary hemochromatosis), iron deficient patients, and iron replete individuals taking oral iron supplements. This proposal will attempt to identify the mechanism by which the human host's iron status and iron supplement use affects the growth and viability of the P. falciparum parasite in red blood cells.

Participants: Healthy adult volunteers, adults with iron deficiency anemia, and patients with hereditary hemochromatosis will be enrolled in this study. Fifteen individuals will be recruited under each of the above three settings. This study involves only subjects over 18 years of age and both males and females will be included.

Procedures (methods): Participation in the study involves undergoing a series of screening tests and donation of blood and either a single time point (for hemochromatosis patients) or a total of three pre-specified time points (for healthy volunteers and those with iron deficiency). The healthy individuals will be asked to take oral iron supplements once daily (325 mg ferrous sulfate) for the duration of this study. Patient's blood will be separated by centrifugation into RBCs and sera, both of which will be used for in vitro studies on the impact of iron status on the growth and viability of Plasmodium falciparum.

ELIGIBILITY:
Inclusion Criteria:

All study participants will need to meet the following eligibility criteria for participation in the study:

1. 18 years of age or older
2. Agree to HIV testing
3. No known malignancy
4. Agree to pregnancy testing (when applicable)
5. Do not have sickle cell disease or trait
6. Do not have thalassemia or thalassemia trait
7. Not taking iron supplementation
8. Have O+ or A+ blood group, and
9. Consent to participate in the study

In addition to the above common study screening tests, additional specific eligibility criteria for the three study groups are as follows:

1. Individuals with iron deficiency:

   Iron deficiency will be diagnosed using the biochemical parameters listed below
   * Serum iron: <40 µg/dL
   * Iron binding capacity (transferrin): <40 µg/dL
   * Saturation (SI/TIBC): <10 percent
   * Hemoglobin: < 9 g/dL
   * Red cell morphology: Hypochromia and microcytosis
   * Plasma or serum ferritin: <10 ng/mL
2. Individuals with Hereditary Hemochromatosis (HH):

   In addition to confirmation with genetic testing, it is expected that patients with HH will have the biochemical parameters listed below. From the genotype standpoint, only patients homozygous for the C282Y and H63D mutations and those that are compound heterozygotes for C282Y/H63D will be enrolled. These are the mutations most associated with iron overload in HH patients. Note that we will have different criteria for men and women. Since women (with and without hemochromatosis) have greater iron losses (secondary to menstruation) in comparison to men, they usually have lower iron stores, lower ferritin levels and lower iron saturation.

   Biochemical parameters:
   * Biochemical markers for patients with HH
   * Serum iron: >65 µg/dL
   * Saturation (SI/TIBC): > 60% men; >50% women
   * Plasma or serum ferritin: >300ng/mL men; >200 ng/mL women

   Each study participant will have been diagnosed (via genetic testing) with HH prior to the enrollment.
3. Healthy volunteers:

Exclusion Criteria:

Patients with HIV, that are pregnant, and those with Sickle cell anemia/trait or Thalassemia/Thal trait will not be eligible to participate in this study as these conditions could interfere with the outcomes of the in vitro studies performed in this proposal.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj Kasthuri, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No